CLINICAL TRIAL: NCT03564977
Title: CD19-targeted CAR-T Cell Therapy for Minimal Residual Disease in B-cell Malignancies After Autologous Stem Cell Transplantation
Brief Title: CD19-targeted CAR-T Cell Therapy for MRD+ B-cell Malignancies After Autologous Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QingdaoCH201805
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Lymphoma, B-Cell; Leukemia, B-Cell; Minimal Disease, Residual
Keywords: CAR-T; minimal residual disease; B cell maliganacy
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-targeted CAR-T cells (Experimental)
  Interventions: Biological: CD19-targeted CAR-T cells

INTERVENTIONS:
Biological: CD19-targeted CAR-T cells — MDR+ patients after autologous stem cell transplantation were treated with CD19-targeted CAR-T cells.

SUMMARY:
The main purpose of this study is to explore the efficacy of CD19-targeted CAR-T cell therapy for minimal residual disease (MRD) in B-cell Malignancies after autologous stem cell transplantation.

DETAILED DESCRIPTION:
Relapse is a common cause of failure in patients with B-cell malignancies after autologous stem cell transplantation. CD19-targeted CAR-T cells showed excellent therapeutic efficiency in B-cell malignancies. Investigators attempt to treat minimal residual disease (MRD)-positive B-cell Malignancies after autologous stem cell transplantation by CD19-targeted CAR-T cells and hope to explore the therapeutic effects of CD19-targeted CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by pathological biopsy in patients with B-cell malignancies and treated by autologous stem cell transplantation.
2. Age 18 to 75 years old, both male and female;
3. Is expected to survive more than 3 months;
4. Physical condition is good: ECOG score≤2;
5. In group of four weeks before Canon imaging examination evaluation body tumor load, recommend line PET - CT examination.
6. General requirements autologous as basic, normal blood T lymphocytes in autologous count must >= 0.2 x10^9 / L;
7. No obvious abnormal heart, liver, kidney, no large wounds that haven't healed on the body;
8. Into groups to participate in voluntarily, good adherence, can cooperate test observation, childbearing age women must be 7 days before starting treatment expert pregnancy test and the results were negative, and signed a written informed consent form.

Exclusion Criteria:

1. Organ failure, such as heart: Class III and IV; liver: to Child grading of liver function grade C; kidney: kidney failure and uremia stage; lung: symptoms of severe respiratory failure; brain: disorder of consciousness;
2. Existing serious acute infection, uncontrollable, or have fester sex and chronic infection, wound in delay no more;
3. Patients with significant graft versus host disease (GVHD) after organ transplant history or allogeneic hematopoietic stem cell transplantation;
4. Systemic autoimmune diseases or immunodeficiency disease, patients with allergic constitution;
5. Coagulation abnormalities and severe thrombosis;
6. Pregnancy and lactation women;
7. Any other chronic disease patients who have been treated with immune agents or hormone therapy;
8. Patients who have participated in other clinical trials or other clinical trials in the past 30 days;
9. The Investigator believe the patients should not participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
Disease control rate | 2 years
Overall survival | 2 years
Progress-free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao, Shandong, China